CLINICAL TRIAL: NCT05956249
Title: Online Cognitive Behavioral Grouptherapy to Improve Depression, Anxiety and Psychological Well-being in Mothers of Babies With Congenital Heart Disease
Brief Title: Online Cognitive Behavioral Groupherapy for Mothers of Babies With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UP 6014/22
Record Dates: First submitted 2023-06-28; First posted 2023-07-21 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2023-06

CONDITIONS: Depressive Symptoms; Anxiety State; Psychological Well-Being
Keywords: Online group therapy; Depression; Anxiety; Well-being; Congenital heart disease
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being; Heart Defects, Congenital | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding will occur for the scientific initiation scholarship holder responsible for reassessing the scales.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Online group therapy (Experimental): Online Cognitive Behavioral grouptherapy for the treatment of depression, anxiety and improvement of emotional well-being.The intervention will be carried out in 6 groups of 6 participants.
  All meetings will be weekly, in groups and will last an average of 1 hour. After the end of the intervention, a scientific initiation fellow will contact the study participants, from both groups, to reapply the scales.
  Interventions: Other: Online group therapy
- Control Group: Without online group therapy (Active Comparator): The control group will only receive the intervention after the reassessment of the scales by the scholarship holder, who is blind to the groups.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Online group therapy — Online group therapy for the treatment of depression, anxiety and improvement of emotional well-being.The intervention will be carried out in 6 groups of 6 participants.
  Arms: Intervention Group: Online group therapy
Other: Control Group — Without intervention at the first moment, but the control group will receive the intervention after the reassessment of the scales by the scholarship holder was done.
  Arms: Control Group: Without online group therapy

SUMMARY:
Introduction: Mothers of babies with congenital heart disease tend to have higher levels of depression, stress and anxiety. Currently, psychological support group technology has been a resource increasingly used by health professionals, with a therapeutic objective as an instrument to promote care. Objective: The aim of this study is to evaluate the effectiveness of a group intervention in improving depression, anxiety and the psychological well-being of mothers of babies with congenital heart disease. Methods: Randomized, parallel clinical trial, in which the factor under study will be online group therapy and the outcome the level of depressive symptoms, anxiety and psychological well-being, assessed using the instruments: BECK-II, BAI and Wellness Scale Ryff's psychological well-being at the beginning and after the intervention. The fellow who will reapply the instruments will be blinded to the groups. Patients will be randomized 1:1, with odd numbers assigned to treatment (online group therapy) and even numbers assigned to controls (no online group therapy). The intervention group will have 8 weekly group consultations, psychoeducational and focused on depression, anxiety and psychological well-being. The sample size was calculated at 36 individuals for each group. Data will be analyzed using the statistical program Statistical Package for Social Sciences (SPSS) version 27.0. For comparison between groups, Student's t test or Kruskall-Wallis or Chi-square test will be used. A two-tailed value of p≤ 0.05 will be considered significant. The normality of instrument scores will be evaluated using the Kolmogorov-Smirnov test. Covariance analysis will be performed to assess the influence of initial scores of anxiety, depression and well-being and their changes after intervention. The effect size will also be calculated. Expected results: It is expected to know and describe the population studied with regard to the level of depressive symptoms, anxiety and psychological well-being. In addition to seeking knowledge about the effectiveness of Group Therapy for these variables.

DETAILED DESCRIPTION:
Design: Randomized, parallel clinical trial, with blinding for the application and evaluation of the instruments.

Participants: 72 mothers (≥ or equal to 18 years old) of babies with congenital heart disease will be included.

Procedures: Patients will be invited to participate in the study on the day of the outpatient consultation or during their children's hospitalization. All participants who agree to participate in the research will respond to the following instruments: BAI, BDI-II and Ryff Psychological Well-Being Scale.

Randomization envelopes will be opened during the interview. Patients in the control group will be informed that they will receive care after the second evaluation.

Patients will be randomized 1:1 according to the order of interviews. Odd numbers assigned to treatment (intervention group therapy) and even numbers assigned to controls. The randomization sequence was generated by the website www.random.org and can be found here: https://www.random.org/sequences/?min=1&max=50&col=1&format=html&rnd=new. Sealed and sequentially numbered envelopes will be made in the order of randomization.

From the randomization, the participants will be allocated to the intervention group (GI) or control group (CG). The intervention will be carried out in 6 groups of 6 participants.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of babies with congenital heart disease, over 18 years of age, assisted at the outpatient clinic or during their child's hospitalization in the pediatric hospitalization or Pediatric ICU of a cardiac hospital who agree to participate and sign the Informed Consent Form.

Exclusion Criteria:

* Mothers unable to answer the questionnaires at the time of application.
* Mothers who do not wish to continue answering the survey.
* Mothers of children over two years old.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Changes in Beck Depression Inventory scores | From baseline to 3 months
  Changes in the depression scores evaluation
Changes in Beck Anxiety Inventory scores | From baseline to 3 months
  Changes in the anxiety scores evaluation

SECONDARY OUTCOMES:
Changes in Ryff psychological well-being scale scores | From baseline to 3 months
  Changes in the well-being scales

CONTACTS AND LOCATIONS:
Overall Officials: MARCIA M SCHMIDT, Principal Investigator — Institute of Cardiology of Rio Grande do Sul
Locations (1):
- Marcia Moura Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No